CLINICAL TRIAL: NCT06241365
Title: The Predictive Role of C-reactive Protein to Albumin Ratio (CAR) in the Treatment of Septic Arthritis in Young Chlidren
Status: Completed | Type: Observational
Sponsor: wangxiaodong (Other)
Responsible Party: Sponsor-Investigator, wangxiaodong, Professor of Medicine, Children's Hospital of Soochow University
Organization: Children's Hospital of Soochow University (Other)
Other Study IDs: 2021KS024
Record Dates: First submitted 2024-01-28; First posted 2024-02-05 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Septic Arthritis
MeSH Terms: conditions — Arthritis, Infectious

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- surgery group: Patients were divided into surgery group and conservative group based on whether the patients underwent surgery.
- conservative group: Patients were divided into surgery group and conservative group based on whether the patients underwent surgery.

SUMMARY:
Purpose: C-reactive protein to albumin ratio (CAR) has emerged as a novel marker of inflammation. However, almost no research has evaluated the role of CAR in septic arthritis (SA). There is currently controversy over the timing of surgery. Our aim is to explore the application of the CAR in predicting the treatment choice for SA in children under 4 years of age.

Methods: Retrospective analysis of the clinical data from children under four years of age admitted to the Department of Orthopedics at Children's Hospital of Soochow University between January 2016 and December 2022 due to SA. Patients were divided into surgery group and conservative group based on whether the patients underwent surgery. The clinical data of the two groups were compared. Multivariate logistic regression analysis was performed to determine the independent predictors for SA requiring surgical intervention. Receiver operating characteristic (ROC) curves were plotted for the independent predictive indicators, and the area under curve (AUC) was determined. The cut-off value was determined using Youden index, and diagnostic accuracy indicators such as sensitivity (SEN), specificity (SPE), positive predictive value (PPV) and negative predictive value (NPV) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* (1) Meeting the aforementioned SA diagnostic criteria, regardless of the affected joint; (2) Completing routine blood and biochemical tests within 24 hours of admission; (3) No surgery or antibiotics administered prior to admission.

Exclusion Criteria:

* (1) Cases of transient synovitis, rheumatism-related diseases (JIA, etc.), simple acute hematogenous osteomyelitis, or acute exacerbation of chronic hematogenous osteomyelitis after revision of the diagnosis; (2) Postoperative iatrogenic infection; (3) Incomplete clinical data.

Ages: 1 Day to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The investigators reviewed the clinical records of patients under 4 years old with SA who were admitted to the Department of Orthopedics at the Children's Hospital of Soochow University for SA treatment between January 2016 and December 2022.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2022-12-18 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
CAR | December 2022
  CAR is an independent predictor indicator for surgery and has good predictive accuracy in chlidren under four years of age with SA.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol